CLINICAL TRIAL: NCT01828554
Title: Pilot Study Evaluating Pharmacokinetic Parameters of Capecitabine Dosing in Patients With Advanced Cancer and Elevated Body Mass Index
Brief Title: Capecitabine Pharmacokinetics(PK)-Actual Versus Ideal Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OS12903; NCI-2013-01267 (Registry Identifier: NCI CTRP); 2013-0280 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2013-04-02; First posted 2013-04-10 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Neoplasms
Keywords: Capecitabine pharmacokinetics PK; Elevated Body Mass Index (BMI); Advanced Solid Tumors
MeSH Terms: conditions — Obesity; Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xeloda (Capecitabine) (Experimental): Cycle 1: Days 1-7 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using "Ideal Body Weight" to calculate dosage. Cycle 1, Day 8-No drug.
  Cycle 1: Days 9-15 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage. Days 16-21-No drug.
  Cycle 2 and greater: Days 1-14 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage.
  Interventions: Drug: Xeloda

INTERVENTIONS:
Drug: Xeloda — Cycle 1: Days 1-7 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using "Ideal Body Weight" to calculate dosage. Cycle 1, Day 8-No drug.
  Cycle 1: Days 9-15 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage. Days 16-21-No drug.
  Cycle 2 and greater: Days 1-14 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage.
  Other Names: Capecitabine

SUMMARY:
The purpose of this research study is to find what happens to capecitabine in the body when dosed using actual versus ideal body weight in subjects with advanced tumors and elevated body mass index.

DETAILED DESCRIPTION:
Cycle 1 : Capecitabine 1,250 mg/m2 orally Per os (PO) once a day (BID) for 7 consecutive days (D1 - D7) will be administered by subject (with Ideal Body Weight being used to determine BSA) for dosage. Day 8-No drug administered.

Capecitabine 1,250 mg/m2 PO BID for 7 more consecutive days (D9 - D15) will be administered by subject (with Actual Body Weight being used to determine BSA) for dosage. There will be 6 consecutive days that no drug will be administered by subject (Days 16-21).

Cycle 2 and beyond: Capecitabine 1,250 mg/m2 PO BID for 14 consecutive days (D1 - D14) will be administered by subject (with Actual Body Weight being used to determine BSA) for dosage. Days 15-21-No drug administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced or metastatic cancer for which capecitabine treatment is considered a standard treatment option.
* Patients with measurable or evaluable disease are eligible
* Patient's Body Mass Index must be 30 kg/m2 or higher.
* Eastern Cooperative Oncology Group performance status 0-2.
* Age >18 years.
* Life expectancy of greater than 12 weeks.
* Patients must have adequate organ and marrow function as defined below:

Hematologic: Absolute Neutrophil Count (ANC) >1000/mcL (microliters), Hemoglobin > 8gm/dL (transfusions permitted) and platelets > 75,000/mcL

Renal: serum creatinine ≤ upper limit of normal (ULN) or creatinine clearance (CrCl) (either estimated or calculated) >60 mL/min/1.73 m for patients with creatinine levels above institutional normal.

Females: Crcl =(140-age)(weight in kg)(0.85)/72 x Serum creatinine

Males: Crcl =(140-age)(weight in kg)/72 x Serum creatinine

Hepatic: Serum Bilirubin ≤ 1.5x ULN and No liver metastases: Aspartate aminotransferase(AST) and Alanine transaminase (ALT) ≤ 2.5x ULN Liver metastases: AST and ALT ≤ 5x ULN

* Ability to understand and the willingness to sign a written informed consent document.
* Capecitabine is contra-indicated in pregnant women because of known detrimental effects on the fetus. A negative pregnancy test is required in all premenopausal women within 14 days of study therapy initiation. Women of child-bearing potential and men with an active female sexual partner must agree to use adequate contraception (hormonal, surgical, barrier methods or abstinence allowed) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who have had systemic chemotherapies or targeted therapies within 3 weeks or radiotherapy within 2 weeks prior to entering the study or those patients whose adverse events from prior therapies have not recovered to < grade 1 and are still considered clinically significant.
* Patients receiving any other investigational agents for cancer treatment.
* Patients with treated, stable brain metastases are allowed to enroll. Patients must be at least 4 weeks from brain radiation and off any medications used to treat brain metastases including steroids. Patients are allowed to be on anti-epileptic medications that are not contraindicated based on the drug-interaction table.
* Patients with any condition of the gastrointestinal tract that is expected to result in an inability to swallow or absorb oral medications (ie. prior surgical procedures affecting absorption and requiring i.v. alimentation). This will be determined at the discretion of the PI.
* Patients may not be taking any concomitant drugs that are contraindicated based on the drug-interaction table.
* Concurrent treatment with warfarin (coumadin) is allowed, but close monitoring of the Prothrombin Time/International Normalized Ratio (PT/INR) is recommended.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active severe infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant or symptomatic cardiac arrhythmia, other malignancies requiring therapy or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women or women who are breastfeeding are excluded from this study because capecitabine is a pregnancy category D drug and is known to pass to the infant in breastmilk.
* Patients with known deficiency of the dihydropyrimidine dehydrogenase (DPD) enzyme.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to capecitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari B. Wisinski, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Xeloda (Capecitabine): Cycle 1: Days 1-7 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using "Ideal Body Weight" to calculate dosage. Cycle 1, Day 8-No drug.
  Cycle 1: Days 9-15 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage. Days 16-21-No drug.
  Cycle 2 and greater: Days 1-14 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage.
  Xeloda: Cycle 1: Days 1-7 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using "Ideal Body Weight" to calculate dosage. Cycle 1, Day 8-No drug.
  Cycle 1: Days 9-15 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage. Days 16-21-No drug.
  Cycle 2 and greater: Days 1-14 (21 day cycle): 1250 mg/m2 Xeloda orally twice a day using Actual Body Weight to calculate dosage.
Period: Overall Study
Arm/Group | Xeloda (Capecitabine)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Xeloda (Capecitabine)
Number analyzed (Participants) | 8
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1
  50-59 years | 2
  60-69 years | 4
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) on Cycle 1 Day 1 and Cycle 1 Day 9
Description: AUC will be calculated for Capecitabine dosed for Ideal Body Weight during the first cycle (days 1-7) and for Capecitabine dosed for Actual Body Weight for first cycle (days 9-15). [nonlinear mixed effects modeling approach]
Time Frame: Up to 15 days
Measure: Mean (Standard Deviation); unit: AUC (ug/ml)*h
Arm/Group | Xeloda (Capecitabine)
Number analyzed (Participants) | 8
AUC (ug/ml)*h
  Cycle 1 Day 1 | 6.84 (7.89)
  Cycle 1 Day 9 | 8.28 (6.64)
Statistical Analysis 1: Comparison: Xeloda (Capecitabine); The null hypothesis that the AUC from cycle 1 day 1 (based on ideal body weight) is equal to the AUC from cycle 1 day 9 (based on actual body weight) was tested against the alternative hypothesis that the AUCs are not equal. A linear mixed effect model with patient specific random effects was conducted; Test type: Other; p = 0.4882, t-test, 2 sided — A paired t-test will be used to compare the PK parameters between the full weight and limited weight based dosing

2. Primary Outcome: Cmax During Cycle 1
Description: Cmax will be reported for Capecitabine dosed for Ideal Body Weight during the first cycle (days 1-7) and for Capecitabine dosed for Actual Body Weight for first cycle (days 9-15). [nonlinear mixed effects modeling approach]
Time Frame: Up to 15 days
Measure: Mean (Standard Deviation); unit: Cmax (ug/ml)
Arm/Group | Xeloda (Capecitabine)
Number analyzed (Participants) | 8
Cmax (ug/ml)
  Cycle 1 Day 1 | 2.44 (1.89)
  Cycle 1 Day 9 | 2.71 (0.98)
Statistical Analysis 1: Comparison: Xeloda (Capecitabine); Test type: Other; p = 0.7497, t-test, 2 sided — A paired t-test will be used to compare the PK parameters between the full weight and limited weight based dosing

3. Secondary Outcome: Response Rate
Description: Responses will be determined using RECIST v. 1.1 criteria and summarized in tabular format. The complete and partial response rates will be calculated and reported along with the corresponding 95% confidence intervals.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Xeloda (Capecitabine)
Number analyzed (Participants) | 8
percentage | 0 [0 to 32.4]

4. Secondary Outcome: Progression Free Survival
Description: Progression-free survival will be analyzed using the Kaplan-Meier method.
Time Frame: Up to 6 months
Population: The median PFS has not been reached (NBR) within the follow-up period of this trial
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Xeloda (Capecitabine)
Number analyzed (Participants) | 8
months | NA [1.4 to NA] — The median Progression Free Survival has (PFS) not been reached (NBR) within the follow-up period of this trial

ADVERSE EVENTS:
Time Frame: up to 9 months
Arm/Group | Xeloda (Capecitabine)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xeloda (Capecitabine) (N=8)
Nausea (Gastrointestinal disorders) | 6 (15)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (8)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (4)
Pain (General disorders) | 2 (3)
Edema limbs (General disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
INR increased (Investigations) | 1 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT01828554/Prot_SAP_000.pdf